CLINICAL TRIAL: NCT04222062
Title: A Randomized Trial Evaluating GLIADEL Compared to Stereotactic Radiosurgery in Subjects With Metastatic Brain Disease
Brief Title: A Study Comparing GLIADEL to Stereotactic Radiosurgery in Metastatic Brain Disease
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Nebraska (Other)
Collaborators: Arbor Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0792-19-FB
Record Dates: First submitted 2020-01-06; First posted 2020-01-09 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Brain Tumor - Metastatic
MeSH Terms: conditions — Brain Neoplasms | interventions — Carmustine; carmustine, poliferprosan 20 drug combination

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized to either 1) the GLIADEL Arm or 2) the Standard of Care Arm (SRS post-op).
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of Care Arm (No Intervention): The tumor will be removed surgically. Within 6 weeks after surgery, the resection will be treated with stereotactic radiosurgery (SRS).
- GLIADEL Arm (Experimental): Once the tumor has been removed, GLIADEL wafers will be applied to the resection cavity. The number of wafers used will be determined by the size of the cavity. Enough wafers should be used so that as much of the cavity is covered as possible.
  Interventions: Drug: Carmustine 7.7Mg Wafer

INTERVENTIONS:
Drug: Carmustine 7.7Mg Wafer — GLIADEL wafers will be placed to cover tumor bed immediately after tumor removal.
  Other Names: GLIADEL
  Arms: GLIADEL Arm

SUMMARY:
This study is being done to see if adding GLIADEL to the site where the tumor was removed works as well as just having the tumor removed with radiation treatment done within six weeks after the surgery to keep the cancer from coming back.

DETAILED DESCRIPTION:
This study is being done to assess the efficacy of GLIADEL, a local chemotherapy, in preventing local recurrence of a metastatic brain tumor compared to stereotactic radiosurgery (SRS) after resection.

100 adult participants with one to four metastatic brain tumors with one tumor needing resection will be enrolled. Participants with prior radiation, lymphoma, small cell, germ cell, unknown primary, or anaplastic thyroid diagnoses will be ineligible. Life expectancy should be greater than 3 months.

Participants will be randomized at the time of surgery to 1) GLIADEL placement at the time of resection or 2) SRS post-operatively to the resection cavity. Any other tumors (up to three) will have SRS as their primary treatment after surgery. SRS will take place within 6 weeks from surgery.

Participants will be evaluated pre-operatively with Magnetic resonance imaging (MRI) brain and neuropsychological testing and will have immediate post-op MRI for extent of resection (EOR) determination. Participants will have SRS to the resection cavity if no GLIADEL was placed and all will have SRS to any other lesions. They will be followed at set intervals to evaluate for local recurrence and neurocognitive changes. The genome of the metastatic brain tumor will be compared to their primary and germline for identification of alterations.

ELIGIBILITY:
Inclusion criteria:

* Age 18 years or older (in states with 18 as age of majority); Age 19 years or older in Nebraska (age of majority)
* Recursive partitioning analysis (RPA) class I, II or III with a Karnofsky Performance Status (KPS) of >/ 60
* Known or suspected primary solid cancer with metastatic brain tumor(s) - up to four in number and up to 4 cm in size with surgical resection planned for at least one site with Gliadel placement planned for only one site
* Laboratory values adequate for patient to undergo surgery safely as determined by the attending neurosurgeon (transfusion permitted to reach goals)
* Women of childbearing potential must have a negative pregnancy test within 7 days of initiating study. (No childbearing potential is defined as age 55 years or older and no menses for two years or any age with surgical removal of the uterus and/or both ovaries)
* Normal coagulation studies (international normalized ratio, INR, ≤ 1.3)
* Estimated survival time of ≥ 3 months (determined by the participant's primary oncologist)
* Participant is willing and able to consent and abide by the protocol

Exclusion criteria:

* Prior treatment to the area of planned resection (surgery, radiation)
* Prior whole brain radiation therapy
* Diagnosis of lymphoma, germ cell cancer, small cell lung cancer, anaplastic thyroid cancer
* Leptomeningeal disease
* Neurodegenerative disorder (e.g. dementia)
* Tumor size > 4 cm
* Karnofsky Performance Status (KPS) < 60
* Inability or unwillingness to co-operate with the requirements of the protocol
* Any other clinically significant medical disease or condition, laboratory abnormality or psychiatric illness that, in the Investigator's opinion, may interfere with protocol adherence or confound efficacy or safety assessment or a subject's ability to give informed consent
* Simultaneous participation in other therapeutic clinical trials
* Severe pulmonary, cardiac or other systemic disease, specifically:

  * New York Heart Association > Grade 2 congestive heart failure within 6 months prior to study entry, unless asymptomatic and well controlled with medication
  * Uncontrolled or significant cardiovascular disease, clinically significant ventricular arrhythmia (such as ventricular tachycardia, ventricular fibrillation, or Torsades des pointes), clinically significant pulmonary disease (such as ≥ Grade 2 dyspnea, according to Common Terminology Criteria for Adverse Events 5.0)
* Participants having any other disease, either metabolic or psychological, which as per Investigator assessment may affect the participant's compliance or place the participant at higher risk of potential treatment complications
* Participant has a bleeding diathesis, or must take anticoagulants, or antiplatelet agents including non-steroidal anti-inflammatory drugs (NSAIDs) at the time of scheduled resection that cannot be stopped for surgery
* Inability to obtain MRI studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-11-06 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Efficacy of GLIADEL compared to Stereotactic Radiosurgery (SRS) | 12 months
  The primary outcome is to evaluate the efficacy of GLIADEL local chemotherapy compared to Stereotactic Radiosurgery (SRS) in preventing local recurrence after resection of a metastatic brain tumor (local recurrence at surgical site).

CONTACTS AND LOCATIONS:
Overall Officials: Michele Aizenberg, MD, Principal Investigator — University of Nebraska
Locations (2):
- United States (2):
  - Henry Ford, Detroit, Michigan
  - University of Nebraska Medical Center, Omaha, Nebraska

IPD SHARING:
Plan to Share IPD: No